CLINICAL TRIAL: NCT06151067
Title: Important Correlation Between Anxiety and Reflux Symptoms in Patients With Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: Evangelic Hospital Kalk Cologne (Other)
Responsible Party: Principal Investigator, Jessica Leers, Prof. Dr. med. Jessica Leers, Evangelic Hospital Kalk Cologne
Other Study IDs: GERD_HADS
Record Dates: First submitted 2023-11-20; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: GERD - Gastro-Esophageal Reflux Disease; Anxiety Disorders
MeSH Terms: conditions — Gastroesophageal Reflux; Anxiety Disorders | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High-Resolution Manometry, Upper-GI endoscopy, pH-Impedance testing — High-Resolution Manometry Upper-GI endoscopy pH-Impedance testing

SUMMARY:
Gastroesophageal reflux disease (GERD) is one of the most common gastroenterological disorders with a reported prevalence of 10% to 20% percent in Europe and the USA and less than 5% in Asia. GERD manifests as heartburn, regurgitation, retrosternal pain, cough, and in some cases dysphagia and holds the possible complication of a Barrett´s esophagus. GERD can appear as non-erosive (NERD) or erosive (ERD). Comorbid symptoms of anxiety and depression are common in GERD patients: The association between anxiety or depression and reflux symptoms has been investigated in previous studies under the aspects of whether existing reflux symptomatology leads to increased anxiety and depression or whether anxiety and depression lead to more severe reflux symptoms. There is a an interaction between GERD and psychosocial disorders.

A long duration of GERD was associated with higher levels of anxiety and depression, and women were more likely to have these symptoms. In patients with Barrett's esophagus, a complication of GERD in which the mucosal cells of the esophagus, under constant exposure to stomach acid, change into a different type of cell normally found in the intestinal tract, rates of anxiety and depression have been reported to be three to five times higher than in the general population.

Anxiety and depression as well as adverse events in life are also independent risk factors for NERD. Patients with NERD show an increased risk for anxiety compared with patients with ERD.

The reporting of somatic symptoms is multifactorial and influenced by psychosocial factors such as socioeconomic status, sex and mental distress. A high somatic symptom load is known to increase anxiety related to health issues, psychological distress and health care utilization. The increased sensation to visceral stimuli in which anxiety and depression play an important role has been discussed as visceral hypersensitivity.

Several studies of patients with reflux symptoms have used the Hopsital Anxiety and Depression Scale (HADS) score as a measure of anxiety and depression and have reported higher anxiety scores than depression scores for this cohort.

The aim of this study was to assess anxiety and depression levels of patients with physiological as well as with pathological DeMeester scores. Further the modulation of anxiety on the severity of reflux symptoms such as fullness, heartburn and dysphagia is examined.

DETAILED DESCRIPTION:
Introduction:

Gastroesophageal reflux disease (GERD) is one of the most common gastroenterological disorders with a reported prevalence of 10% to 20% percent in Europe and the USA and less than 5% in Asia. GERD manifests as heartburn, regurgitation, retrosternal pain, cough, and in some cases dysphagia and holds the possible complication of a Barrett´s esophagus. GERD can appear as non-erosive (NERD) or erosive (ERD). In the diagnosis of the reflux disease the DeMeester score is used as a measure of esophageal acid exposure time. Important differential diagnosis are benign functional disorders of the esophagus such as is functional heartburn or functional dysphagia. Comorbid symptoms of anxiety and depression are common: The association between anxiety or depression and reflux symptoms has been investigated in previous studies under the aspects of whether existing reflux symptomatology leads to increased anxiety and depression or whether anxiety and depression lead to more severe reflux symptoms. The results are inconsistent: In younger patients (18 - 40 years) with gastroesophageal reflux disease (GERD) the prevalence of anxiety and depression is higher than in those without GERD. There is an independent association between GERD, anxiety and current depression. Patients with anxiety are more likely to experience GERD symptoms and these symptoms seem to be more severe in anxious patients. Anxiety and depression intensify symptom perception. Patients with GERD have a higher incidence of anxiety, depression and sleep disturbances than those without GERD, and there is an association between psychosocial disorders and an increased risk of anxiety. Thus, there is a an interaction between GERD and psychosocial disorders, which has been discussed as the "psychoemotional effects of GERD". GERD is considered to be an independent source of stress.

A long duration of GERD was associated with higher levels of anxiety and depression, and women were more likely to have these symptoms. In patients with Barrett's esophagus, a complication of GERD in which the mucosal cells of the esophagus, under constant exposure to stomach acid, change into a different type of cell normally found in the intestinal tract, rates of anxiety and depression have been reported to be three to five times higher than in the general population.

Anxiety and depression as well as adverse events in life are also independent risk factors for NERD. Patients with NERD show an increased risk for anxiety compared with patients with ERD.

The reporting of somatic symptoms is multifactorial and influenced by psychosocial factors such as socioeconomic status, sex and mental distress. A high somatic symptom load is known to increase anxiety related to health issues, psychological distress and health care utilization. The increased sensation to visceral stimuli in which anxiety and depression play an important role has been discussed as visceral hypersensitivity.

Several studies of patients with reflux symptoms have used the Hopsital Anxiety and Depression Scale (HADS) score as a measure of anxiety and depression and have reported higher anxiety scores than depression scores for this cohort.

The aim of this study was to assess anxiety and depression levels of patients with physiological as well as with pathological DeMeester scores. Furthermore, the modulation of anxiety on the severity of reflux symptoms such as fullness, heartburn and dysphagia is examined.

2. Methods Statement of ethics The present study was conducted according to Declaration of Helsinki principles and was approved by the Ethics Committee of the Medical Faculty of the University of Cologne. All patients provided their online informed consent. The study has not been registered in any study register.

Study design We conducted a prospective observational cohort study with one measurement time on admission.

Participants We enrolled all patients who were referred to the "Reflux and swallowing problems center" of the Clinic for General and Visceral Surgery of the University Hospital Cologne, Germany, between January 2020 and July 2021. Only patients were included for analysis who completed the HADS-D. All patients underwent gastrointestinal function diagnostics with esophagogastroduodenoscopy, 24-hour pH-metry, high-resolution manometry and esophagography. Psychometric data were collected using the HADS. The criteria for indication for surgery were positive DMS, presence of hiatal hernia, changes in the esophagus due to reflux such as Barrett esophagus or inflammation, poor tolerance of medication, low level of symptom control through medication and lifestyle, decreased quality of life, long duration of the disease and substantial comorbidities. Not all criteria needed to be fullfied.

Questionnaires We used the HADS in its German version for assessing anxiety (HADS-A) and depression levels (HADS-D). Self-report is used to assess the severity of anxious and depressive symptoms during the past week, which is recorded on two subscales with seven items each, each item ranging from 0 - 3, adding up to a maximal total score of 21. For both subscales a cutoff score for caseness of > 8 is recommended (27).

Data analysis In evaluating the HADS scores we labeled scores on the subscales of HADS-A of 8 and over 8 as "anxious" and those on the subscale of HADS-D of 8 and over 8 as "depressed". We differentiated between mildly (HADS score on the subscale 8-10), moderately (HADS 11 - 14) and severely (HADS 15 - 21) anxious or depressed.

The DMS was determined using 24h pH impedance testing which included the following values in the score: percentage of time with esophageal pH < 4 of the total measurement period, percentage of time with pH < 4 during the waking phase (upright position), percentage of time with pH < 4 during sleep phase (supine position), total number of reflux episodes during the measurement period, number of reflux episodes with duration > 5 min, duration of the longest reflux episode.

In evaluating the DMS we labeled scores as negative (physiological) (< 14.72) or positive (pathological) (> 14.72). The positive scores were differentiated into mild (14.72 - 30), moderate (30 - 80) and severe (<80).

Statistical Analysis Statistical analysis was performed using IBM SPSS Statistics. Continuous variables were presented as mean and standard deviation, categorical data as frequencies with percentages. To identify differences between two groups, an independent samples T-test was performed for parametric data, whereas a Mann-Whitney U test was performed for non-parametric data. Furthermore, a Chi-square test for independence or Fischer's Exact test respectively was performed in case of categorical data. Correlation between parameters was investigated using Pearson correlation coefficient for parametric data and Spearman correlation coefficient for non-parametric data. A p-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of reflux who present at the consultation hour at the department of General, Visceral, Tumor and Transplantation Surgery of the University Hospital of Cologne
* Patients who underwent Upper GI Endoscopy, High-Resolution Manometry and pH-Impedance testing who completed the HADS questionnaire were included into the study.

Exclusion Criteria:

* Patients without knowledge of the German language
* Patients who did not complete the HADS questionnaire
* Patients who did not complete all diagnostic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of reflux (heartburn, regurgitation, retrosternal pain) who present at the consultation hour at the department of General, Visceral, Tumor and Transplantation Surgery of the University Hospital of Cologne were included into the study. All patients underwent Upper GI Endoscopy, High-Resolution Manometry and pH-Impedance testing who completed the HADS questionnaire were included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression | During diagnostic workup of patients with gastroesophageal reflux disease as baseline characteristics
  Anxiety and depression are evaluated during diagnostic workup of patients using the HADS questionnaire. In evaluating the HADS scores were grouped into subscales of HADS-A of =8 and >8 as "anxious" and those on the subscale of HADS-D of 8 and over 8 as "depressed". It is differentiated between mildly (HADS score on the subscale 8-10), moderately (HADS 11 - 14) and severely (HADS 15 - 21) anxious or depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Leers, Prof., Principal Investigator — Department of Functional Upper GI Surgery
Locations (1):
- Department of General, Visceral, Tumor and Transplantation Surgery, University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided